CLINICAL TRIAL: NCT02652156
Title: Transversus Abdominis Plane (TAP) Block Study for Postoperative Pain Control
Brief Title: TAP Block for Postoperative Pain Control
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Operational barriers at the site.
Sponsor: Joshua Herskovic (Other)
Responsible Party: Sponsor-Investigator, Joshua Herskovic, Anesthesiologist, Midwestern Regional Medical Center
Organization: Midwestern Regional Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MZ2014035
Record Dates: First submitted 2015-11-19; First posted 2016-01-11 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Pain, Postoperative
Keywords: transversus abdominis plane; postoperative; pain
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Bupivacaine; Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Single Injection of Bupivacaine (Active Comparator): Subjects will undergo post-operative pain relief treatment with a single injection of Bupivacaine, a local anesthetic injected into the transversus abdominis plane.
  Interventions: Drug: Bupivacaine
- Single Injection of Exparel® (Active Comparator): Subjects will undergo post-operative pain relief treatment with a single injection of Exparel®, a liposomal form of bupivacaine, into the transversus abdominis plane
  Interventions: Drug: Exparel®
- Continuous infusion of Ropivacaine (Active Comparator): Subjects will be treated with a continuous infusion of the local anesthetic Ropivacaine with the ON-Q® pump
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Bupivacaine — 60 ml Bupivacaine 0.25% will be drawn via 60 ml Syringe. The syringe will be connected and a 10ml flush syringe containing 10ml 0.9% Normal Saline (NS) will be connected to the end of an IV extension set via a 3-way stopcock and Luer lock connections. The Bupivacaine 0.25% syringe will be connected to the stopcock. The distal end of the IV connection will be connected to the injection needle. The entire setup will be flushed with 0.9% NS via flush syringe. The TAP space will also be located under ultrasound guidance and verified by using the 0.9% NS flush syringe. Once in the TAP space, 30 ml Bupivacaine 0.25% will be injected into the TAP space. This dose will be decreased to 25 ml for patients under 70 kg. The process will be repeated on the opposite side TAP block.
  Other Names: Marcaine; Sensorcaine
  Arms: Single Injection of Bupivacaine
Drug: Exparel® — 20 ml Exparel (266 mg) will be drawn into a 20 ml syringe. A 20 ml Bupivacaine 0.25% syringe and the syringe containing the Exparel solution will be connected to the end of an IV extension set via a 3-way stopcock. The IV connection will be connected to the injection needle. The setup will be flushed with the Bupivacaine syringe. The TAP space will be located under ultrasound guidance. 133mg of Exparel will be injected into the TAP space. After injection, the syringe will be exchanged for the Bupivacaine syringe and 20ml Bupivacaine injected into the space. The process will be repeated on the opposite side TAP block.
  Other Names: bupivacaine liposome injectable suspension
  Arms: Single Injection of Exparel®
Drug: Ropivacaine — 40 ml Bupivacaine 0.25% will be drawn via two 20ml Syringes. A Bupivacaine 20ml syringe will be connected to an IV extension via a 3-way stopcock and Luer lock. The IV will be connected to an injection tuohy needle and flushed with NS. The TAP space will be located using ultrasound guidance. 15 ml Bupivacaine 0.25% will be injected. A catheter will be threaded through the tuohy needle into the TAP space. 5ml Bupivacaine 0.25% will then be injected. The catheter will be secured via standard technique. The process will be repeated for the opposite side. Patients will receive a filled ON-Q system. The ON-Q system contains Ropivacaine 0.2%. The pump will run at 7 ml/hr. per side.
  Other Names: Naropin
  Arms: Continuous infusion of Ropivacaine

SUMMARY:
This clinical trial will examine differences in the effectiveness between three (3) commonly used methods and/or medications used to perform a transversus abdominis plane (TAP) block for post-operative pain control. The transversus abdominis muscle is either side between the lowest rib and the hip bone. Group A subjects will undergo post-operative pain relief treatment with a single injection of Bupivacaine injected into the TAP. Group B subjects will undergo post-operative pain relief treatment with a single injection of Exparel®, a liposomal form of bupivacaine into the TAP. Group C subjects will be treated with a continuous infusion of the local anesthetic ropivacaine with the ON-Q® pump. There will be no placebo group in this study.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give written informed consent
* Scheduled for open abdominal surgery
* American Society of Anesthesiologists physical status 1 to 3

Exclusion Criteria:

* Inability to understand the study or provide written informed consent
* Inability to follow protocol instructions
* Complicated history of chronic opioid use including daily use of opioids for a period greater than 2 weeks prior to surgery
* Allergy to local anesthetic agents
* Contraindication to regional nerve block such as:
* Bleeding disorder
* Sepsis
* Infection at site of block
* Body Mass Index (BMI) >40
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2016-04-16 (Actual); Study Completion 2016-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Herskovic, MD, Principal Investigator — Midwestern Regional Medical Center

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Injection of Bupivacaine | Single Injection of Exparel® | Continuous Infusion of Ropivacaine
Started | 4 | 6 | 4
Completed | 3 | 6 | 4
Not Completed | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Injection of Bupivacaine | Single Injection of Exparel® | Continuous Infusion of Ropivacaine | Total
Number analyzed (Participants) | 4 | 6 | 4 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 4 | 12
  >=65 years | 0 | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 3 | 9
  Male | 2 | 2 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 5 | 4 | 13
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 2 | 6
  White | 1 | 4 | 2 | 7
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 6 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: Total Dosage of Narcotic
Description: The total use of analgesic medications will be recorded during the 3 days immediately following surgery.
Time Frame: 3 postoperative days
Population: 1 patient in the Continuous Infusion of Ropivacaine group required no narcotics immediately following surgery (recovery room) due to continuing effect of the blockade. Patients are removed from study upon discharge in later postoperative days.
Measure: Mean (Standard Deviation); unit: Mophine Equivalent Units
Arm/Group | Single Injection of Bupivacaine | Single Injection of Exparel® | Continuous Infusion of Ropivacaine
Number analyzed (Participants) | 3 | 6 | 4
Mophine Equivalent Units
  Narcotic Use - Day of Surgery - Recovery room: number analyzed (Participants) | 3 | 6 | 3
  Narcotic Use - Day of Surgery - Recovery room | 23.2 (19.1) | 14.4 (11.8) | 35.7 (22.6)
  Narcotic Use - Postoperative Day 0 | 33.0 (34.0) | 42.2 (39.9) | 45.0 (23.9)
  Narcotic Use - Postoperative Day 1 | 87.7 (106.5) | 139.0 (194.6) | 47.9 (36.4)
  Narcotic Use - Postoperative Day 2: number analyzed (Participants) | 2 | 6 | 3
  Narcotic Use - Postoperative Day 2 | 127.0 (61.0) | 103.3 (112.7) | 44.7 (36.4)
  Narcotic Use - Postoperative Day 3: number analyzed (Participants) | 1 | 4 | 1
  Narcotic Use - Postoperative Day 3 | 318.0 (0) | 41.6 (40.6) | 68.0 (0)

2. Secondary Outcome: Postoperative Vomiting (Events)
Description: Total number of vomiting episodes over the three postoperative days.
Time Frame: 3 postoperative days
Population: No vomiting events were reported by any study subjects.
Measure: Number; unit: Vomiting Events
Arm/Group | Single Injection of Bupivacaine | Single Injection of Exparel® | Continuous Infusion of Ropivacaine
Number analyzed (Participants) | 3 | 6 | 4
Vomiting Events | 0 | 0 | 0

3. Secondary Outcome: Patient Reported Pain by VAS Scale
Description: Patients will rate their pain by VAS scale 1 day post surgery. Scale is a 0 to 10 visual analog scale with 0 representing no pain and 10 representing severe pain.
Time Frame: Postoperative Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Injection of Bupivacaine | Single Injection of Exparel® | Continuous Infusion of Ropivacaine
Number analyzed (Participants) | 3 | 6 | 4
score on a scale | 4.4 (0.4) | 3.8 (0.9) | 4.5 (0.4)

4. Secondary Outcome: Patient Reported Pain by VAS Scale
Description: Patients will rate their pain by VAS scale 2 days post surgery. Scale is a 0 to 10 visual analog scale with 0 representing no pain and 10 representing severe pain.
Time Frame: Postoperative Day 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Injection of Bupivacaine | Single Injection of Exparel® | Continuous Infusion of Ropivacaine
Number analyzed (Participants) | 3 | 6 | 4
score on a scale | 4.2 (1.6) | 2.0 (1.2) | 5.3 (1.9)

5. Secondary Outcome: Patient Reported Pain by VAS Scale
Description: Patients will rate their pain by VAS scale 3 days post surgery. Scale is a 0 to 10 visual analog scale with 0 representing no pain and 10 representing severe pain.
Time Frame: Postoperative Day 3
Population: Two patients in each of the Single Injection of Bupivacaine and Continuous Infusion of Ropivacaine groups were discharged prior to post-operative day 3. Pain rating data for these subjects were not collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Injection of Bupivacaine | Single Injection of Exparel® | Continuous Infusion of Ropivacaine
Number analyzed (Participants) | 1 | 6 | 2
score on a scale | 4.0 (0) | 2.2 (1.2) | 3.8 (0.8)

6. Secondary Outcome: Number of Days Required for a Patient to Get Out of Bed
Description: Patients will be assessed each day following the day of surgery for the ability to get out of bed.
Time Frame: Assessed daily for up to 3 days post-surgery
Population: All 3 patients in the Single Injection of Bupivacaine cohort required 1 day to be able to get out of bed.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Single Injection of Bupivacaine | Single Injection of Exparel® | Continuous Infusion of Ropivacaine
Number analyzed (Participants) | 3 | 6 | 4
days | 1.0 (0.0) | 0.8 (0.4) | 0.3 (0.5)

7. Secondary Outcome: Number of Days Required for a Patient to Walk Unassisted
Description: Patients will be assessed each day following the day of surgery for the ability to walk unassisted
Time Frame: Assessed daily for up to 3 days post-surgery
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Single Injection of Bupivacaine | Single Injection of Exparel® | Continuous Infusion of Ropivacaine
Number analyzed (Participants) | 3 | 6 | 4
days | 1.3 (0.5) | 1.5 (0.5) | 1.3 (0.5)

ADVERSE EVENTS:
Time Frame: 4 Days
Arm/Group | Single Injection of Bupivacaine | Single Injection of Exparel® | Continuous Infusion of Ropivacaine
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/6 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT02652156/Prot_SAP_000.pdf